CLINICAL TRIAL: NCT05246202
Title: Latinx Hazardous Drinkers With Clinical Anxiety: Effectiveness Trial of a Personalized Normative Feedback Intervention
Brief Title: Personalized Feedback Intervention for Latinx Drinkers With Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Distinguished Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003237; 1R01AA029807-01 (NIH)
Record Dates: First submitted 2021-11-29; First posted 2022-02-18 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Abuse; Anxiety
Keywords: Latinx; Hispanic; Personalized Feedback Intervention
MeSH Terms: conditions — Alcoholism; Anxiety Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anxiety-alcohol personalized feedback intervention (AA-PFI 2.0) (Experimental): Participants complete the brief (~20-30 minute) AA-PFI 2.0 at baseline.
  Interventions: Behavioral: Alcohol-Anxiety Personalized Feedback Intervention 2.0
- Control personalized feedback intervention (C-PFI) (Active Comparator): Participants complete the brief (~20-30 minute) C-PFI at baseline.
  Interventions: Behavioral: Control Personalized Feedback Intervention

INTERVENTIONS:
Behavioral: Alcohol-Anxiety Personalized Feedback Intervention 2.0 — AA-PFI 2.0 is a culturally adapted, brief, computer-delivered, personalized feedback intervention to address alcohol misuse in the context of clinical anxiety.
  Other Names: AA-PFI 2.0
  Arms: Anxiety-alcohol personalized feedback intervention (AA-PFI 2.0)
Behavioral: Control Personalized Feedback Intervention — C-PFI is a brief, computer-delivered, personalized feedback intervention on exercise and nutrition.
  Other Names: C-PFI
  Arms: Control personalized feedback intervention (C-PFI)

SUMMARY:
The purpose of this study is to develop, evaluate the acceptability/feasibility (Phase IA), and test (Phase IB) the effectiveness of a brief, integrated, single-session, computer-based, culturally adapted personalized feedback intervention (PFI) designed to enhance knowledge regarding adverse anxiety-alcohol interrelations, increase motivation and intention to reduce hazardous drinking, and reduce positive attitudes and intention regarding anxiety-related alcohol use among Latinx hazardous drinkers with anxiety.

DETAILED DESCRIPTION:
In the first phase, the investigators will collect qualitative and quantitative feedback from focus groups to refine intervention content and evaluate treatment acceptability and feasibility of a novel, brief, integrated, culturally adapted computer-based personalized feedback intervention (PFI). In the second phase, Latinx hazardous drinkers with clinical anxiety will be recruited and randomly assigned to either the refined culturally adapted anxiety-alcohol PFI (AA-PFI 2.0) or a control PFI (C-PFI). Initial screening will be conducted via telephone; baseline and post-treatment data will be collected in-person; and 1-, 3-, and 6-month follow-up data will be collected online remotely.

ELIGIBILITY:
Inclusion Criteria:

* Being between the age of 21 to 75 years of age
* Being self-identified as Latinx or Hispanic
* Fluent in Spanish
* Meeting criteria for current hazardous drinking pattern
* Meeting criteria for clinical anxiety
* Being able to provide written, informed consent

Exclusion Criteria:

* Being involved in alcohol or other substance use program
* Currently pregnant
* Current engagement in psychotherapy for anxiety

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Motivation to Reduce Alcohol Consumption Scale | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The 1-item Motivation to Reduce Alcohol Consumption Scale will be used to measure current motivation/intention to reduce alcohol. Participants will be asked to select the statement that best describes their motivation/intention to reduce drinking (e.g., "I really want to cut down on drinking alcohol and intend to in the next month"). Higher scores on this measure indicate greater motivation/intention to reduce alcohol consumption (possible range (0-7).
Modified Drinking Motives Questionnaire-Revised | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The Modified Drinking Motives Questionnaire-Revised will be used to assess expectancies of drinking. For the current study, the 4-item "Coping-anxiety" subscale will be used as a measure of expectancies of drinking to reduce/cope with anxiety. The measure utilizes a 5-point Likert scale ranging from 1 (almost never/never) to 5 (almost always/always). Scores are averaged with higher scores indicating greater expectancies of drinking to reduce/cope with anxiety (possible range 1 to 5).
Alcohol Attitudes Scale | Change from Baseline Pre PFI completion to Baseline Post PFI completion
  The 7-item Alcohol Attitudes Scale will be utilized to measure maladaptive attitudes for drinking (e.g., "Drinking alcohol is good"). Items are rated on a Likert-type scale from 1 (strongly disagree) to 7 (strongly agree). Scores will be averaged to create a composite score (possible range 1 to 7). Higher scores indicate greater maladaptive attitudes for drinking.

SECONDARY OUTCOMES:
Overall Anxiety Severity and Impairment Scale | Change from Baseline Pre PFI Completion to 6-months Post PFI Completion
  The 5-item Overall Anxiety Severity and Impairment Scale will be used to assess anxiety symptom severity and impairment. Each of the items is rated on a Likert-type scale ranging from 0 to 4. Items are summed to produce a total score (possible range 0 to 20).
Alcohol Use Disorders Identification Test | Change from Baseline Pre PFI Completion to 6-months Post PFI Completion
  The Alcohol Use Disorders Identification Test will be used to assess drinking quantity, craving, and related consequences to alcohol use. The 10 items are rated with various Likert-type scales. The measure produces a total score by adding all of the items of the measure with higher scores indicating greater problems with alcohol (possible range 0 to 40).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Zvolensky, Ph.D., Principal Investigator — University of Houston
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Treatment Outcomes, and Racial Equity, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.